CLINICAL TRIAL: NCT00112034
Title: A Multi-Center, Randomized, Blinded, Parallel-Group Study of AVONEX Compared With AVONEX in Combination With Oral Methotrexate, Intravenous Methylprednisolone, or Both in Subjects With Relapsing Remitting MS Who Have Breakthrough Disease on AVONEX Monotherapy.
Brief Title: AVONEX® Combination Trial - "ACT"
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Dennis Cunningham, Associate Director, Medical Affairs, Biogen Idec
Allocation: Randomized | Model: Factorial | Masking: Double
Other Study IDs: C-865
Record Dates: First submitted 2005-05-27; First posted 2005-05-30 (Estimated); Last update posted 2008-05-09 (Estimated); Status verified 2008-05

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple Sclerosis; Relapsing-Remitting; AVONEX; Combination; Methotrexate; IV Methylprednisolone; IVMP; ACT; MTX
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Methotrexate; Methylprednisolone

INTERVENTIONS:
Drug: Methotrexate
Drug: IV methylprednisolone

SUMMARY:
The purpose of this study is to determine the efficacy and safety of combination therapy with AVONEX plus low dose oral methotrexate (MTX), every other month courses of intravenous methylprednisolone (IVMP), or both in patients with continued disease activity on AVONEX monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 55, inclusive
* Diagnosis of MS
* A relapsing-remitting course
* Expanded Disability Status Scale (EDSS) score 0.0-5.5 inclusive at Baseline
* Currently receiving AVONEX® therapy
* Treated with AVONEX® for at least 6 consecutive months prior
* Breakthrough disease (clinical relapse or gadolinium-enhancing MRI lesion) during the prior 12 months, at least 6 months after initiating AVONEX therapy.

Exclusion Criteria:

* History of cirrhosis, chronic hepatitis, or currently active hepatitis
* History of poorly-controlled hypertension, diabetes mellitus, or peptic ulcer disease
* History of aseptic bone necrosis, osteoporosis, or osteoporosis-related bone fracture
* History of steroid-induced psychosis.
* History of or abnormal laboratory results indicating significant illness
* History of severe allergic or anaphylactic reactions or known drug hypersensitivity or intolerance to MTX, IVMP, or AVONEX®.
* History of allergy to albumin
* History of any episode of suicidal ideation or severe depression within 3 months of the Screening Visit.
* History of seizure within 3 months prior to the Screening Visit.
* Diagnosis of primary progressive, secondary progressive, or progressive relapsing MS
* MS relapse with onset within 60 days prior to the Baseline Visit
* Any metallic or electronic material or device in the body, or condition that precludes the subject from undergoing MRI with gadolinium administration
* A clinically significant infectious illness (e.g., cellulitis, abscess, pneumonia, septicemia) within 30 days of the Screening Visit
* Abnormal blood tests, performed at the Screening Visit, which exceed any of the limits defined by the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 350
Dates: Start 2003-06; Primary Completion 2006-06 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Brain MRI lesion activity measured by the combined number of T2-hyperintense lesions at Month 12 that are new or enlarged since Baseline
effectiveness of AVONEX® and IVMP plus MTX in trying to reduce lesion activity on brain MRI

SECONDARY OUTCOMES:
Gadolinium enhancing lesion number on brain MRI, relapse rate, MS Functional Composite change, whole brain atrophy progression

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A. Cohen, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- MS Academic Coordinating Center, Cleveland, Ohio, United States